CLINICAL TRIAL: NCT04413695
Title: Lung Ultrasound as a Point of Care Test for Living Donor Liver Transplant Recipients: A Prospective Observational Study
Brief Title: Lung Ultrasound as a Point of Care Test for Living Donor Liver Transplant Recipients.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Principal Investigator, Gaurav Sindwani, Assistant Professor, Institute of Liver and Biliary Sciences, India
Other Study IDs: ILBSIndia 2
Record Dates: First submitted 2020-05-30; First posted 2020-06-04 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-10

CONDITIONS: Liver Transplant; Complications
Keywords: liver transplant; lung ultrasound; chest x ray

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Liver transplant is now a standard treatment for end-stage liver disease patients. Pulmonary complications are common in the perioperative period and are associated with adverse outcomes. This includes atelectasis, pneumothorax, pleural effusion, pulmonary edema, and collapse. Risk factors for the same are extensive surgery, transfusion of blood products, fluid overload, hemodynamic instability, coagulation abnormalities, renal dysfunction, and reperfusion syndrome. CXR with clinical judgment plays a key role in diagnosing pulmonary complications. However diagnostic ability of CXR is limited and moreover it is associated with unnecessary radiation exposure. Recently, lung USG has come up as an easily available tool to detect peri-op pulmonary complications. The technique is very easy to perform, less time-consuming, and totally cost-effective. Moreover, it can be easily learned by clinicians with a standard level of ability to handle an ultrasound probe for abdominal scans. In the setting of geriatric and ICU patients, fragility and immobility have a strong impact on the quality of a chest radiograph. So, the routine application of lung USG in this setting may significantly improve the outcome. Multiple studies have suggested that Lung USG is superior to CXR in diagnosing these lung conditions. Hence, this study aims to compare the lung ultrasound with CXR in detecting perioperative pulmonary complications in patients undergoing live donor liver transplantation.

DETAILED DESCRIPTION:
This is a prospective observational study on liver transplant recipient patients, until postoperative day seven. After approval of the ethical committee and written informed consent, all liver transplant recipients meeting inclusion criteria are enrolled in the study. Patient characteristics like the cause of liver failure, CTP scoring, MELD Na scoring, graft vs recipient weight ratio, age, weight, height, BMI, pulmonary and other comorbidities are noted. Both lung ultrasound and CXR are done simultaneously in all patients on: one day prior to surgery and post-operatively from day 1 to day 7. Ultrasound is done by an experienced anesthesiologist with good experience in lung ultrasound, while the CXR was interpreted by the another physician. Based on the findings in the different regions of the thorax, a lung ultrasound score (LUS) is calculated as the following:- Each hemithorax is divided into anterior-lateral sectors (from parasternal to posterior axillary lines) and posterior sectors (from posterior axillary to paravertebral line). Each sector then divided into upper and lower halves taking the third intercostal space as reference, so that 4 areas could be finally identified for each hemithorax. The probe was set perpendicular, oblique, and parallel to the ribs to assess the degree of lung aeration with a total of 8 zones to be examined using a linear and convex probe. Image interpretation will be according to Lung Ultrasound Score. Lung ultrasound score varies from 0-3 [0 = normal aeration; 1 = moderate loss of aeration (interstitial syndrome, defined by multiple spaced B lines, or localized pulmonary edema, defined by coalescent B lines in less than 50% of the intercostal space examined in the transversal plane, or subpleural consolidations); 2 = severe loss of aeration (alveolar edema, defined by diffused coalescent B lines occupying the whole intercostal space); 3 = complete loss of lung aeration (lung consolidation defined as a tissue pattern with or without air bronchogram)]. The LUS is calculated as the sum of the 12 regional scores. Along with the LUS, other complications like atelectasis, pulmonary edema, consolidation, effusion and collapse are also noted. The LUS will be correlated with clinically relevant perioperative pulmonary complications (POPC) and the length of the ICU stay. The clinically relevant POPC are defined when any of the following present:

1.Increase in RR >25/min 2. The need of FIO2>10% 3. Increase Need of PS by 5cm of H2O and need of PEEP by 2cm of H20 4.The need of IMV, reinitiation of NIV, and insertion of ICD. Both CXR and lung ultrasound findings are compared with respect to the day of appearance of complications on CXR and ultrasound. In addition the data will be collected for the total duration of the complication, total length of icu and hospital stay.

.

ELIGIBILITY:
Inclusion Criteria:

Age 18 to 65yrs All end stage liver disease patients undergoing live donor liver transplantation

Exclusion Criteria:

Patients not giving consent for enrollment Any structural cardiac condition Dead donor liver transplant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: End stage liver disease patients
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-11-11 (Actual); Primary Completion 2021-09-25 (Estimated); Study Completion 2021-09-25 (Estimated)

PRIMARY OUTCOMES:
Comparison of day of appearance of pulmonary complications on ultrasound and chest Xray | till post operative seventh day
  Comparison of day of appearance of pulmonary complications on ultrasound and chest Xray

SECONDARY OUTCOMES:
Incidence and types of postoperative pulmonary complications after live donor related liver transplant (LDLT) | First post-operative seven days
  Incidence and types of postoperative pulmonary complications after live donor related liver transplant (LDLT)
Correlation of lung ultrasound score with clinically relevant perioperative pulmonary complications and length of icu stay | First post-operative seven days
  Correlation of lung ultrasound score with clinically relevant perioperative pulmonary complications and length of icu stay

CONTACTS AND LOCATIONS:
Overall Officials: gaurav sindwani, md, Study Chair — ilbs
Locations (1):
- Gaurav Sindwani, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Feltracco P, Carollo C, Barbieri S, Pettenuzzo T, Ori C. Early respiratory complications after liver transplantation. World J Gastroenterol. 2013 Dec 28;19(48):9271-81. doi: 10.3748/wjg.v19.i48.9271. PMID 24409054
- [Background] Ruchonnet-Metrailler I, Blanchon S, Luthold S, Wildhaber BE, Rimensberger PC, Barazzone-Argiroffo C, Mc Lin VA. Pulmonary complications after liver transplantation in children: risk factors and impact on early post-operative morbidity. Pediatr Transplant. 2018 Jul 17:e13243. doi: 10.1111/petr.13243. Online ahead of print. PMID 30019517
- [Background] Tierney DM, Boland LL, Overgaard JD, Huelster JS, Jorgenson A, Normington JP, Melamed RR. Pulmonary ultrasound scoring system for intubated critically ill patients and its association with clinical metrics and mortality: A prospective cohort study. J Clin Ultrasound. 2018 Jan;46(1):14-22. doi: 10.1002/jcu.22526. Epub 2017 Oct 6. PMID 28984373
- [Background] Zhao Z, Jiang L, Xi X, Jiang Q, Zhu B, Wang M, Xing J, Zhang D. Prognostic value of extravascular lung water assessed with lung ultrasound score by chest sonography in patients with acute respiratory distress syndrome. BMC Pulm Med. 2015 Aug 23;15:98. doi: 10.1186/s12890-015-0091-2. PMID 26298866
- [Result] Yin W, Zou T, Qin Y, Yang J, Li Y, Zeng X, Kang Y; Chinese Critical Ultrasound Study Group (CCUSG). Poor lung ultrasound score in shock patients admitted to the ICU is associated with worse outcome. BMC Pulm Med. 2019 Jan 3;19(1):1. doi: 10.1186/s12890-018-0755-9. PMID 30606165
- [Result] Soummer A, Perbet S, Brisson H, Arbelot C, Constantin JM, Lu Q, Rouby JJ; Lung Ultrasound Study Group. Ultrasound assessment of lung aeration loss during a successful weaning trial predicts postextubation distress*. Crit Care Med. 2012 Jul;40(7):2064-72. doi: 10.1097/CCM.0b013e31824e68ae. PMID 22584759